CLINICAL TRIAL: NCT04700631
Title: Extracellular Vesicles as Biomarkers for Chronic Renal Failure
Acronym: VE-IRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0104
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Renal Failure; Urinary Extracellular Vesicle
Keywords: urinary extracellular vesicle; Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy subject (Active Comparator): healthy subjects : no medical history, in particular cardiovascular, without drug treatment, without proteinuria, normal BMI
  Interventions: Diagnostic Test: urinary extracellular vesicle concentration; Diagnostic Test: blood sample
- CRF patients (Experimental): CRF patients : eGFR estimated according to the MRDR formula less than 89 mL/min/1,73m²
  Interventions: Diagnostic Test: urinary extracellular vesicle concentration; Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: urinary extracellular vesicle concentration — urinary extracellular vesicle concentration will be determined in urine samples from CRF and healthy patients
Diagnostic Test: blood sample — blood sample in order to determine creatin level

SUMMARY:
The recent discovery of extracellular vesicles (EV) as a mechanism of intercellular communication has made it possible to develop a new field of health research and could bring new information on the pathological mechanisms of renal diseases. Definition of physiologic and pathologic values of urinary extracellular vesicles (EVu) between healthy subjects and chronic kidney diseases (CKD) patients could be a new tool for follow up of renal diseases. EV are found in all biological fluids including urine, that's why they are increasingly analyzed in renal pathologies. The main objective of this study is to determine the physiological values and the pathological thresholds of EVu.

ELIGIBILITY:
Inclusion Criteria:

* subject > 18 years old
* healthy subjects : no medical history, in particular cardiovascular, without drug treatment, without proteinuria, normal BMI
* CRF patients : eGFR estimated according to the MRDR formula less than 89 mL/min/1,73m²

Exclusion Criteria:

* patients under dialysis protocols
* renal transplant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
variation of urinary extracellular vesicle concentration between both groups | one day
  variation of urinary extracellular vesicle concentration between both groups : healthy and CRF patients Urinary extracellular vesicle concentrations will be measured as number of extracellular vesicles per mL of urine

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacob V, de Berny Q, Brazier F, Presne C, Lion J, Ouled-Haddou H, Metzinger-Le Meuth V, Choukroun G, Metzinger L, Guillaume N. Quantification of Urine and Plasma Levels of Extracellular Vesicles in a Cohort of Kidney Transplant Recipients and Chronic Kidney Disease Patients. Int J Mol Sci. 2025 Apr 11;26(8):3635. doi: 10.3390/ijms26083635. PMID 40332150